CLINICAL TRIAL: NCT06316934
Title: The Use of Lavender Aromatherapy to Decrease Women's Anxiety and Perception of Pain During Office Hysteroscopy Procedure
Brief Title: Lavender Aromatherapy to Decrease Anxiety/Pain Perception During Office Hysteroscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: IRB202302181
Record Dates: First submitted 2024-02-06; First posted 2024-03-19 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Anxiety; Pain, Procedural
Keywords: Aromatherapy; Hysteroscopy; Lavender
MeSH Terms: conditions — Anxiety Disorders; Pain, Procedural

STUDY DESIGN:
Intervention Model Description: The participants will be randomized into two arms - aromatherapy or placebo. The protocol will be the same for the two arms except that the towel held over the mouth will be scented either with lavender essential oil or distilled water. The clinic nurse will prepare the scented towel and hand it to the participant according to the random assignment.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization will be performed once the patient agrees to participate and has signed the consent document. A random number generator will be used to designate each arm of the study. Odd numbers will be assigned to the aromatherapy arm while the even numbers will be assigned to the placebo arm. Each assignment will be placed into a sealed opaque numbered enveloped. After the participant has agreed to participate, the clinic nurse will open the envelope to identify the study arm.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Prior to starting the procedure, the clinic nurse will prepare the distilled water on a paper towel by applying two drops of each solution on a paper towel. The patients will hold the paper towel over their nose and then they will be asked to take two deep breaths. Before the physician comes in, the nurse will ask the participant to take a deep breath while holding the towel 3 inches from her face and will instruct the participant to continue to take normal breaths subsequently
  Interventions: Other: Placebo
- Experimental (Experimental): Prior to starting the procedure, the clinic nurse will prepare the aromatherapy Lavender essential oil on a paper towel by applying two drops of each solution on a paper towel. The patients will hold the paper towel over their nose and then they will be asked to take two deep breaths. Before the physician comes in, the nurse will ask the participant to take a deep breath while holding the towel 3 inches from her face and will instruct the participant to continue to take normal breaths subsequently
  Interventions: Drug: Lavandula angustifolia, Aura Cacia

INTERVENTIONS:
Drug: Lavandula angustifolia, Aura Cacia — Lavender essential oil will be placed on paper towel which patient will deeply inhale prior to the start of the procedure.
  Arms: Experimental
Other: Placebo — Distilled water will be placed on paper towel which patient will deeply inhale prior to the start of the procedure.
  Other Names: Distilled water
  Arms: Placebo

SUMMARY:
Office hysteroscopy is an invaluable practice to treat a myriad of gynecological processes. However, a limiting factor is the perceived pain and anxiety. In a randomized pilot study, treatment with lavender aromatherapy will significantly decrease the stress/anxiety levels associated with office hysteroscopy, as measured on a visual analogue scale and the Hospital Anxiety and Depression Scale (HADS) questionnaire when compared to control subjects receiving distilled water placebo.

DETAILED DESCRIPTION:
This study is a randomized placebo control trial. The designation of aromatherapy versus placebo will be randomized, but no procedures will be performed for study purposes that would not be normally performed for a patient's clinical assessment.

Women scheduled for Office Hysteroscopy at the Women's Health Medical Plaza Clinic (UF Shands) clinic will be invited to participate. Participants who meet inclusion criteria will be randomized to the aromatherapy or the placebo group after informed consent is obtained and immediately before undergoing the Hysteroscopy procedure. Sequentially numbered sealed opaque envelopes containing the identity of the study arm will be used for randomization. The Medical Plaza clinic nurse will prepare the aromatherapy versus distilled water on the paper towel with two drops of each utilized. Before the physician comes in, the nurse will ask the participant to take a deep breath while holding the towel 3 inches from her face and will instruct the participant to continue to take normal breaths subsequently. It will not be possible to blind the participants or the examiner to the assigned group since the lavender oil will have a different scent than the placebo. However, the use of distilled water on the towel will allow the possibility that the deep breathing accompanying the instruction may have an effect on reported pain and anxiety.

Vaginoscopy approach will be utilized to perform the procedure. This avoids the use of a speculum in the vagina or tenaculum to grasp the cervix. This is a atraumatic technique that reduces pain stimuli generated from the cervix and the vagina when using manipulating instruments. Vaginoscopy relies on hydrodilation of the cervical canal for entry of a small-caliber scope. This technique involves distending the vaginal vault with normal saline and advancing the scope to the posterior fornix. Gently pulling back until the external cervical os is visualized and then the scope is advanced into the cervical canal.

The participant will undergo the standard clinic exam in a standardized order. The participants will complete the Hospital Anxiety and Depression Survey (HADS) at baseline. The HADS (Appendix II) is a reliable instrument for detecting states of depression and anxiety in the setting of a hospital medical outpatient clinic; it is available in English and Spanish versions. This will be used to establish their baseline anxiety levels. Participants will then be asked to rate their level of anxiety and pain immediately before beginning the exam, immediately after hysteroscope placement, and 15 min after termination of the study using a 10-point visual analogue scale and the Wong-Baker pain scale. At the end, the participants will also be asked to rate their satisfaction with the visit overall on a visual analogue scale.

ELIGIBILITY:
* Inclusion Criteria:

  * Women aged 18 and over
  * Scheduled to undergo office hysteroscopy procedure
  * Able to give informed consent
  * Able to read and write in English
  * Anxiety score > 0 on a numerical scale at baseline
* Exclusion Criteria:

  * Any contraindication to office hysteroscopy (active pelvic infection, confirmed cervical or endometrial cancer severe hypertension, or any other condition that might be worsened by an uncomfortable test)
  * Allergy to lavender oil, or any of its components
* Withdrawal Criteria

  * The patient requests terminating participation

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-04-21 (Actual); Study Completion 2025-04-21 (Actual)

PRIMARY OUTCOMES:
Determine the change in pain scores from baseline to immediate post-procedure. | 30 minutes
  Participants will then be asked to rate their level of pain immediately before beginning the exam, immediately after catheter placement, and 15 min after termination of the study using the Wong-Baker pain scale. 0 would be no pain at all and 10 would be the worst pain.
Determine change in anxiety scores from baseline to immediate post-procedure. | 30 minutes
  Participants will then be asked to rate their level of anxiety immediately before beginning the exam, immediately after catheter placement, and 15 min after termination of the study using a 10-point visual analog scale. 0 corresponds with a pleasant face and represents no anxiety at all and 10 corresponds with a face in distress and represents high levels of anxiety.
Determine level of satisfaction after the procedure | 5 minutes
  At the end, the participants will also be asked to rate their satisfaction with the visit overall on a Likert scale. If patient's are satisfied they would choose "Strongly Agree" and if they are dissatisfied with the experience they can choose "Strongly disagree." Agree, disagree and neutral would be the additional choices.

CONTACTS AND LOCATIONS:
Overall Officials: Tiffani-Amber Miller, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data is not intended to be shared with other researchers

REFERENCES:
- [Background] Buzzaccarini G, Alonso Pacheco L, Vitagliano A, Haimovich S, Chiantera V, Torok P, Vitale SG, Lagana AS, Carugno J. Pain Management during Office Hysteroscopy: An Evidence-Based Approach. Medicina (Kaunas). 2022 Aug 20;58(8):1132. doi: 10.3390/medicina58081132. PMID 36013599
- [Background] Fouks Y, Kern G, Cohen A, Reicher L, Shapira Z, Many A, Yogev Y, Rattan G. A virtual reality system for pain and anxiety management during outpatient hysteroscopy-A randomized control trial. Eur J Pain. 2022 Mar;26(3):600-609. doi: 10.1002/ejp.1882. Epub 2021 Nov 23. PMID 34748679
- [Background] Gambadauro P, Navaratnarajah R, Carli V. Anxiety at outpatient hysteroscopy. Gynecol Surg. 2015;12(3):189-196. doi: 10.1007/s10397-015-0895-3. Epub 2015 May 13. PMID 26283891
- [Background] Vitale SG, Caruso S, Ciebiera M, Torok P, Tesarik J, Vilos GA, Cholkeri-Singh A, Gulino FA, Kamath MS, Cianci A. Management of anxiety and pain perception in women undergoing office hysteroscopy: a systematic review. Arch Gynecol Obstet. 2020 Apr;301(4):885-894. doi: 10.1007/s00404-020-05460-2. Epub 2020 Mar 5. PMID 32140807